CLINICAL TRIAL: NCT00979446
Title: Developing a Multi-Domain Intervention to Maintain Cognitive Health in Sedentary Adults Ages 60 - 80
Brief Title: Passport to Brain Wellness in Sedentary Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Responsible Party: Brian C. Martinson, PhD, Senior Research Investigator, HealthPartners Research Foundation
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 03-024S2; 3R01AG023410-05S2 (NIH)
Record Dates: First submitted 2009-09-16; First posted 2009-09-18 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Mild Cognitive Impairment; Alzheimer's Disease
Keywords: Interactive phone-based intervention with written materials; Older adults; Physical activity; Cognitive stimulation; Social engagement
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Guided (Experimental)
  Interventions: Behavioral: Guided
- Self-directed (Active Comparator)
  Interventions: Behavioral: Self-directed

INTERVENTIONS:
Behavioral: Guided — Engaged in a 4 month pilot of a multi-domain lifestyle intervention with a phone coach
  Arms: Guided
Behavioral: Self-directed — Received study materials but no phone coaching
  Arms: Self-directed

SUMMARY:
Numerous modifiable lifestyle factors have been identified that may affect the risk of older adults developing mild cognitive impairment (MCI) and Alzheimer's disease (AD). Evidence suggests that interventions to reduce risk factors and enhance protective factors would be beneficial in slowing cognitive decline and decreasing the risk of incident MCI and AD. The overall objective of this pilot study, funded as a supplement to Keep Active Minnesota (KAM) (03-024; R01-AG023410) is to develop and test the feasibility of conducting a multi-domain intervention to maintain cognitive health in adults ages 60-80 with the goal of reducing the incidence of and slowing progression to MCI and other more severe forms of cognitive decline.

DETAILED DESCRIPTION:
The initial aim of the project was to recruit 20 cognitively intact adults ages 60-80 from one health plan, assessing them at baseline with respect to their cognitive health, multiple lifestyle factors, biomarkers and biometrics, engaging them in a 12 week lifestyle intervention and re-assessing them immediately post-intervention.

Specific Aims

1. Design a multi-domain, lifestyle intervention to increase PA, social integration and cognitive stimulation, and improve nutrition in sedentary, cognitively intact adults, age 60 to 80.
2. Assess the feasibility of implementing such a multi-domain intervention:

   1. recruit and screen 20 sedentary, cognitively intact adults aged 60 to 80 from a health plan,
   2. obtain baseline measures of cognitive function, physical and social activities, mood, nutrition, height and weight, vascular risk factors of blood pressure and fasting lipids, and biomarkers of inflammation,
   3. engage these adults in a 4 month pilot of this multi-domain lifestyle intervention with a phone coach and
   4. obtain post-intervention measures of cognitive functioning, physical and social activities, mood, nutrition, vascular risk factors of blood pressure and fasting lipids, and biomarkers of inflammation.

After successfully recruiting the first 20 subjects, we determined that the grant budget would allow us to enrich the study by recruiting 40 more subjects. A second, comparison arm was added. The first study arm received the intervention as described above. Subjects assigned (by chance) to the comparison arm received study materials but did not have a phone coach assigned. The additional 40 subjects were genotyped with respect to the apolipoprotein E4 (apoE4) allele.

This feasibility pilot of an evidence-based intervention targets protective lifestyle factors related to cognitive health, including physical and social activities, cognitive stimulation and nutrition. The information gained on intervention design, implementation, and subject recruitment, will guide development of a full-scale intervention study of primary prevention of cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the ages of 60 and 80
* Have had HealthPartners insurance for 11 out of the 12 months prior to recruitment
* Engage in less than 90 minutes per week of moderate intensity physical activity
* Works or volunteers 20 hours total per week or less
* Telephone Interview for Cognitive Status (TICS) score of 31 and above

Exclusion Criteria:

* Modified Charlson scores >=3 (calculated using prior year diagnoses)
* Nonskin cancer
* Congestive heart failure
* Coronary heart disease
* Psychotic Illness
* Substance abuse
* Terminal illness

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2008-06; Primary Completion 2009-05 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
We will use this pilot to determine the feasibility of carrying out a full-scale randomized trial to test the efficacy of our intervention. | Six months after the baseline visit

CONTACTS AND LOCATIONS:
Overall Officials: Brian C Martinson, PhD, Principal Investigator — HealthPartners Institute
Locations (1):
- HealthPartners Research Foundation, Bloomington, Minnesota, United States